CLINICAL TRIAL: NCT01146821
Title: Multi-centre, Open-label, Phase II Clinical Trial for Determination of the Optimal Dose of Fish Oil in Patients With Severe Sepsis
Brief Title: Fish OIL Optimal dosE Determination Study
Acronym: FOILED
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Low enrollment/ expiration of the grant
Sponsor: University Hospital Carl Gustav Carus (Other)
Collaborators: University of Giessen (Other); Clinical Evaluation Research Unit at Kingston General Hospital (Other); GWT-TUD GmbH (Other)
Responsible Party: Principal Investigator, Axel R. Heller, MD, University Hospital Carl Gustav Carus
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FK-FOILED; 2010-021018-49 (EudraCT Number)
Record Dates: First submitted 2010-06-17; First posted 2010-06-22 (Estimated); Last update posted 2017-04-19 (Actual); Status verified 2017-04

CONDITIONS: Sepsis
MeSH Terms: conditions — Sepsis | interventions — fish oil triglycerides

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Standard care (No Intervention): Standard care
- standard care + 0.20gm/kg fish oil (Active Comparator): standard care + 0.20gm/kg fish oil
  Interventions: Dietary Supplement: 0.20 gm/kg fish oil
- standard care + 0.50 gm/kg fish oil (Active Comparator): standard care + 0.50 gm/kg fish oil
  Interventions: Dietary Supplement: 0.50 gm/kg fish oil

INTERVENTIONS:
Dietary Supplement: 0.20 gm/kg fish oil — Group 2: 7 patients will receive 0.20gm/kg of ideal body weight [IBW] fish oil in addition to standard care
  Other Names: Omegaven
  Arms: standard care + 0.20gm/kg fish oil
Dietary Supplement: 0.50 gm/kg fish oil — Group 3: 7 patients will receive 0.50 gm/kg of ideal body weight [IBW] fish oil in addition to standard care.
  Other Names: Omegaven
  Arms: standard care + 0.50 gm/kg fish oil

SUMMARY:
The primary objective of this trial is to determine the safety and efficacy of IV fish oil doses of 0.20 g/kg and 0.50 g/kg, compared to a control group, in critically ill patients with severe sepsis by examining organ function, blood safety and biochemical parameters, markers of systemic inflammation and innate immunological parameters

DETAILED DESCRIPTION:
Objectives: The overall objective is to determine the effect of IV fish oil on 28-day mortality of critically ill patients with severe sepsis. However, prior to such a large trial, we need to determine the optimal dose of IV fish oils in this population. Therefore, the primary objective of this proposal (FOILED) is to determine the safety and efficacy of IV fish oil doses of 0.20 g/kg and 0.50 g/kg, compared to a control group, in critically ill patients with severe sepsis by examining organ function, blood safety and biochemical parameters, markers of systemic inflammation and innate immunological parameters.

Study Design: This is a multi-centre, open-label, phase I dose ranging clinical trial with prospective controls.

Setting: 2 tertiary care ICUs in Germany (Universitätsklinikum Carl Gustav Carus, Dresden and University Hospital Giessen and Marburg, Giessen).

Patients: Mechanically ventilated adult patients (>18 years old) admitted to ICU with clinical evidence of sepsis, sepsis associated organ dysfunction, and high expression of inflammatory cytokines.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients
* Requiring invasive or non-invasive ventilation
* Clinical evidence of sepsis
* Presence of one or more organ failures

Exclusion Criteria:

* >24 hours from admission to ICU to time of consent
* Low level of inflammatory cytokine (IL-6(qualitative assay <100 pg/ml)
* lack of commitment to full aggressive care (anticipated withholding or withdrawing treatments in the first week)
* Immunocompromised (post-organ transplantation, HIV, neutropenic [<1000 PMN], steroids >20 mgs/day for 6 months).
* Chronic non-invasive ventilation (except if they become mechanically ventilated)
* Platelet count of < 30 GPt/L
* Pregnant patients. Urine/blood tests for pregnancy will be done on all women of childbearing age by each site as part of standard of ICU practice.
* Previous enrollment in this study
* Enrollment in other ICU intervention study
* Allergy to fish or fish oil (shellfish allergy not an exclusion criterion)
* Has already received enteral or IV omega-3 fatty acids during this hospitalization and current ICU admission.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2013-10; Primary Completion 2017-04 (Actual); Study Completion 2017-04 (Actual)

PRIMARY OUTCOMES:
Change in SOFA score | Day 1-10
  As the primary goal of this study is to establish the safety of high doses of IV fish oils, our primary outcomes will be change in SOFA score (organ function) and biochemical parameters of safety (i.e. blood lipid levels, coagulation parameters, bleeding episodes, standard biochemistry).

SECONDARY OUTCOMES:
Markers of systemic inflammation | Day 1-10
  Our secondary outcomes include markers of systemic inflammation [pro-calcitonin [PCT], C-reactive protein [CRP], interleukin-1 [IL-6] and IL-10) and markers of innate immunity [such as lipopolysaccharide [LPS] ex-vivo stimulation of tumor necrosis factor-alpha [TNF-α]].
Clinical outcomes | Day 1-28
  In addition, we plan to collect clinical outcomes such as ICU and hospital length of stay, number of infections, length of ventilation, and ICU, 28-day, and hospital mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Axel R. Heller, MD, Principal Investigator — University Hospital Dresden, Germany; Daren Heyland, MD, PhD, Study Chair — Kingston General Hospital, Canada; Rupinder Dhaliwal, RD, Study Director — Kingston General Hospital, Canada
Locations (2):
- Germany (2):
  - University Hospital Dresden, Dresden
  - University Hospital Giessen and Marburg, Giessen

REFERENCES:
- [Background] Pradelli L, Mayer K, Muscaritoli M, Heller AR. n-3 fatty acid-enriched parenteral nutrition regimens in elective surgical and ICU patients: a meta-analysis. Crit Care. 2012 Oct 4;16(5):R184. doi: 10.1186/cc11668. PMID 23036226
- [Background] Heller AR, Rossler S, Litz RJ, Stehr SN, Heller SC, Koch R, Koch T. Omega-3 fatty acids improve the diagnosis-related clinical outcome. Crit Care Med. 2006 Apr;34(4):972-9. doi: 10.1097/01.CCM.0000206309.83570.45. PMID 16484909
- [Background] Heller AR, Rossel T, Gottschlich B, Tiebel O, Menschikowski M, Litz RJ, Zimmermann T, Koch T. Omega-3 fatty acids improve liver and pancreas function in postoperative cancer patients. Int J Cancer. 2004 Sep 10;111(4):611-6. doi: 10.1002/ijc.20291. PMID 15239141
- [Background] Heller AR, Fischer S, Rossel T, Geiger S, Siegert G, Ragaller M, Zimmermann T, Koch T. Impact of n-3 fatty acid supplemented parenteral nutrition on haemostasis patterns after major abdominal surgery. Br J Nutr. 2002 Jan;87 Suppl 1:S95-101. doi: 10.1079/bjn2001462. PMID 11895160
- [Background] Mayer K, Fegbeutel C, Hattar K, Sibelius U, Kramer HJ, Heuer KU, Temmesfeld-Wollbruck B, Gokorsch S, Grimminger F, Seeger W. Omega-3 vs. omega-6 lipid emulsions exert differential influence on neutrophils in septic shock patients: impact on plasma fatty acids and lipid mediator generation. Intensive Care Med. 2003 Sep;29(9):1472-81. doi: 10.1007/s00134-003-1900-2. Epub 2003 Jul 25. PMID 12897994
- [Background] Manzanares W, Dhaliwal R, Jurewitsch B, Stapleton RD, Jeejeebhoy KN, Heyland DK. Parenteral fish oil lipid emulsions in the critically ill: a systematic review and meta-analysis. JPEN J Parenter Enteral Nutr. 2014 Jan;38(1):20-8. doi: 10.1177/0148607113486006. Epub 2013 Apr 22. PMID 23609773
- [Background] Pradelli L, Eandi M, Povero M, Mayer K, Muscaritoli M, Heller AR, Fries-Schaffner E. Cost-effectiveness of omega-3 fatty acid supplements in parenteral nutrition therapy in hospitals: a discrete event simulation model. Clin Nutr. 2014 Oct;33(5):785-92. doi: 10.1016/j.clnu.2013.11.016. Epub 2013 Dec 4. PMID 24345520